CLINICAL TRIAL: NCT05555472
Title: The Effectiveness of the Youth Initiated Mentoring Approach for Juvenile Delinquents
Brief Title: The Youth Initiated Mentoring Approach for Juvenile Delinquents
Status: Unknown | Phase: Not Applicable | Type: Interventional
Last Known Status: Recruiting
Sponsor: University of Amsterdam (Other)
Collaborators: ZonMw: The Netherlands Organisation for Health Research and Development (Other); YIM Foundation Netherlands (JIMwerkt.nl) (Unknown); Halt (Halt.nl) (Unknown)
Responsible Party: Principal Investigator, Levi van Dam, Study Principal Investigator, University of Amsterdam
Allocation: Non-Randomized | Model: Parallel | Masking: None | Purpose: Prevention
Other Study IDs: ZonMw #744130101
Record Dates: First submitted 2022-09-07; First posted 2022-09-27 (Actual); Last update posted 2022-09-27 (Actual); Status verified 2022-09

CONDITIONS: Juvenile Delinquency; Youth Initiated Mentoring (YIM) Approach
Keywords: Natural mentoring; Youth Initiated Mentoring; Delinquency; Juvenile; Adolescents; Prevention; Reoffending

STUDY DESIGN:
Intervention Model Description: Youths will be non-randomly allocated to either a YIM trained Halt professional (N = 31), or a Halt professional not trained in the YIM approach (N = 31). These professionals will implement the Halt-plus-YIM-condition (N =150) or the CAU Halt-condition (N = 150), respectively. Random allocation of cases to Halt professionals was not possible because Halt's distribution office considers individuals' workload. Despite non-random allocation, conditions will be comparable in terms of (1) the professionals who deliver the intervention (i.e., same educational level and from the same region), and (2) case type and severity. Allocation of a youths' case to a professional, is independent of type of offense and its severity as well as the evaluation of number of risk factors present in youth. In addition, due to the equal number of professionals per region, similar distributions of youths per region are expected.
Masking Description: Participants are aware of following the Halt-intervention (with a YIM) but they are not aware of the existence of the other condition. Adolescents in the CAU Halt-condition are not aware of participants following the Halt-YIM condition (and possibly not aware of the YIM approach itself) and vice versa.
  The care providers, YIM trained and non-trained professionals, can only include participants for either the experimental or control condition respectively. Whether the adolescent is a participant, only becomes known if the professional explicitly asks the adolescent. After their invitation, adolescents are redirected to give their consent. Actual registration of participants is registered by the researchers. Researchers do not actively communicate which adolescents have registered for the study.
  Both the investigator and outcomes assessor are aware of which participant is in which condition but are not directly involved with the participants nor the procedure in the conditions.
Oversight: Data Monitoring Committee: No | FDA-regulated Drug: No | FDA-regulated Device: No

ARMS (2):
- Care-as-usual Halt-condition (Active Comparator): Participants in this arm will follow the regular Halt-intervention. Halt professionals, not trained in YIM-approach, will be instructed to follow their regular working procedure. On average, the intervention consists of 3 meetings: an initial meeting, an intervention meeting, and a closing meeting. The aim is to complete the intervention within 100 days (min.-max.: 1-6 meetings, 1-20 hours). During the initial meeting, compulsory activities are screening and risk assessment, reflection on the committed offense/crime, and parental involvement. Based on these activities, the duration and the content of the intervention are determined. Professionals can select activities from 5 different modules: (1) reflection on behaviour, (2) parental involvement, (3) social skills training, (4) victim-offender reconciliation, and (5) future. A form of victim-offender reconciliation, however, is compulsory. Professionals are required to register relevant information regarding the Halt-process.
  Interventions: Behavioral: Halt-intervention
- Halt-plus-YIM-condition (Experimental): Participants in this arm will follow the Halt-plus-YIM-intervention. YIM trained Halt professionals implement the YIM approach in their regular working procedure in 7 steps: (1) during risk assessment, they support youth in identifying a YIM; (2) during the course of the study, professionals will be instructed to motivate and explain the YIM approach in cases with 3 or more meetings; (3) if a YIM is nominated, a meeting between the professional and the YIM takes place; (4) to 'position' the YIM, a joint meeting is arranged to discuss expectations/goals of all involved parties; (5) interim contact between professional and YIM takes place; (6) a joint evaluative meeting takes place; (7) if agreed upon, closure of Halt's engagement takes place. Note, the YIM often remains involved after this completion. Professionals register on the Halt- and YIM-process and whether the approach was deployed: 'NO' (i.e., only step 1), 'PARTLY' (i.e., steps 1 and 2) or 'YES' (i.e., at least step 3 or 4).
  Interventions: Behavioral: Halt-intervention; Behavioral: Youth Initiated Mentoring (YIM) approach

INTERVENTIONS:
Behavioral: Halt-intervention — The main aim of the Halt-intervention is to reduce the risk for reoffending. Seven sub-goals are implemented to work towards this main aim: (1) youths gain insight in (the consequences of) their behaviour; (2) strengthening youths' social skills; (3) youths are able take responsibility for the consequences of their behaviour; (4) victim-offender reconciliation; (5) youths are able to access support from own social network and, if necessary, access to formal support; (6) parents gain insight their child's behaviour; and (7) if youths complete the intervention, they do not receive a registration on their criminal record. With a compulsory screening and risk assessment at the start of the intervention, it is determined which sub-goals fit the adolescents' needs. The intervention gives Halt professionals the opportunity to identify adolescents (and families) in vulnerable circumstances and to guide them towards formal support, like youth care organisations or addiction treatment centres.
Behavioral: Youth Initiated Mentoring (YIM) approach — The YIM approach focuses on strengthening naturally existing relationships between youth and non-parental adults within their own social network (Van Dam & Schwartz, 2020). It stems from the idea "it takes a village to raise a child (Educational Civil Society)", which implies that other adults are co-responsible for the development of youth in their environment (Bowers et al., 2015). The YIM approach can be implemented in a formal context; expertise from the own social network is then combined with expertise from professionals (Van Dam & Verhulst, 2018). Professionals support youth in identifying and positioning a "YIM" as part of a broader intervention (Van Dam & Schwartz, 2020). Youths are responsible for asking their YIM and once agreed upon, the YIM is "positioned". The YIM offers advice/support and plays a role during the intervention followed by the youth. Youth, parents, YIMs and professionals work together to set expectations and goals for the engagement of the YIM.
  Arms: Halt-plus-YIM-condition

SUMMARY:
Natural or informal mentorship could potentially be considered effective in preventing or reducing delinquent behaviour. In the Youth Initiated Mentoring (YIM) approach, youths are supported by professionals in identifying and nominating a natural mentor within their own social network. The approach focuses on strengthening these naturally existing relationships with non-parental adults. Until now, little (quasi-)experimental research is conducted on the YIM approach. In the Netherlands, juvenile offenders between 12-18 years are referred to Halt, where they are required to follow a tailored intervention with the aim of preventing reoffending and increasing youths' future opportunities. Since 2019, the YIM approach is implemented as part of the Halt-intervention. The researchers will examine whether the YIM approach is an effective addition to the Halt-intervention. More specifically, whether it contributes to (1) strengthening youths' resilience, (2) decreasing or halting the need for formal support, and (3) decreasing or halting the development of juvenile delinquency.

This quasi-experimental trial aims to include 300 youths referred to Halt. Youths will be non-randomly allocated to either a YIM trained Halt professional (N = 31), or a Halt professional not trained in the YIM approach (N = 31). These professionals will implement the Halt-plus-YIM-condition (N =150) or the care-as-usual Halt-condition (N = 150), respectively. Random allocation of youth cases to Halt professionals was not possible because Halt's distribution office considers individuals' workload. Despite non-random allocation, conditions will be comparable in terms of (1) the professionals who deliver the intervention (i.e., same educational level and from the same region), and (2) case type and severity (i.e., allocation is independent of type of offense and its severity as well as the evaluation of number of risk factors present in youth). Researchers will perform a multi-informant measurement strategy. Youths are our primary informants, but parents of youths are also approached to participate. Youth and parent questionnaires related to several youth and family outcomes will be administered at baseline, 100 days after baseline (post-test), and nine months after baseline (follow-up). Researchers will also collect information registered by Halt professionals in Halt's registration system. Read detailed description for more information on outcomes.

DETAILED DESCRIPTION:
Main aims and hypotheses

The main aim is to examine whether the YIM approach is an effective addition to the Halt-intervention. More specifically, researchers will examine whether the addition of a YIM to the Halt-intervention contributes to (1) strengthening adolescents' resilience (by stimulating protective factors), (2) decreasing or halting the need for formal support and (3) decreasing or halting the development of juvenile delinquency.

H1: It is expected that the YIM approach will strengthen youth resilience:

1. Improvement in social network quality as indexed by increased perceived social support, perceived mattering, and relatedness to others;
2. Improvement of social skills as indexed by increased social resourcefulness;
3. Increased feelings of autonomy and competence;
4. Decreased positive attitudes towards delinquency;
5. Stronger commitment to the social environment as indexed by increased school attachment, and structured free-time activities;
6. Stronger commitment to the social environment by increased school performance, school attachment and structured free-time activities.

H2: It is expected that YIM contributes to halting or decreasing the need for (formal) support.

H3: It is expected hat YIM contributes to halting or decreasing self-reported delinquency.

H4: It is expected that hypotheses three and four are mediated by an increase in resilience factors, such as perceived mattering, self-determination, and social control.

H5: It is expected that the effects of the YIM approach will work better for some than for others, therefore moderators such as demographic factors, psychosocial problems, mentor relationship quality, peer network quality, parental monitoring, and treatment characteristics (i.e., Halt-intervention characteristics and YIM approach characteristics) will be explored.

In addition, for parents the presence of a YIM could lead to an increase in family resilience, perceived social support and social resourcefulness, and a decrease in parental stress and need for (formal) support. It is also expected that they report less delinquent behaviour in their child.

Abovementioned youth and parent outcomes will be assessed as outcome measures, but exploratively also included in mediator analysis. Check measurements at "outcomes".

Methods/Design

Design

This quasi-experimental study was designed in co-creation with Halt professionals, policy officers and Halt management. Multiple design- and brainstorm sessions took place during the first phase of the study. Researchers presented several frameworks/ideas based on theory, which were then further developed, selected, combined, or adjusted together with Halt professionals. One part of the co-creation process was related to designing the participant flow of the study-to align this in an optimal way with the Halt working process. Several research steps (informed consent, pre-test, post-test, follow-up measurement, etc.) were printed on smaller post-its, which were then, in smaller groups, rearranged, organised, and pasted in an overview of the Halt working process. Ideas of the different groups were combined, strengths and pitfalls were assessed, and the most feasible design was selected. Another part of the co-creation process related to the selection of outcome measures. In a brainstorm session with Halt professionals, professionals selected outcome cards (i.e., change in which outcomes were expected after following the Halt-intervention and which after following the Halt-YIM intervention). In several adjacent brainstorm sessions about Halt's 'Theory of Change' with Halt policy officers and management, the outcome domains of Halt were further specified. Both the 'Theory of Change' discussion and the outcome cards discussion, then served as input for the researchers in the selection of outcome measures. These co-creation processes are in line with the Q-sort technique.

The study sample will consist of N = 300 Dutch adolescents (12-18 years) referred to Halt by a prosecutor, the police, a special investigating civil servant or a school attendance civil servant after committing an offense or crime. Common offenses are public inebriation, nuisance, and violation of the compulsory education law, common crimes are theft and vandalism. Adolescents will be non-randomly allocated to either a YIM trained Halt professional (N = 31) or a Halt professional not trained in the YIM approach (N = 31). These professionals will implement the Halt-plus-YIM-condition (N =150) or the care-as-usual (CAU) Halt-condition (N = 150), respectively. Despite non-random allocation to the Halt-plus-YIM and CAU, conditions will be comparable in terms of (1) the professionals who deliver the intervention and (2) case type and severity (see brief summary).

Researchers will perform a multi-informant measurement strategy. Youths are the primary informants, but parents of youths in both conditions are also approached to participate. Both youths and parents fill out questionnaires at baseline, 100 days after baseline (post-test) and nine months after baseline (follow-up). Participants with shortened cases (with less than three meetings) are excluded from post-test and follow-up measurements. Access is granted to relevant information about youth registered by Halt professionals in Halt's registration system.

Participant recruitment

Participants will be recruited by Halt professionals; data collection will be organised by the researchers. YIM-trained professionals will be responsible for recruiting participants for the Halt-YIM-condition (N = 150), non-trained Halt professionals will be responsible for recruiting participants for the CAU Halt-condition (N = 150). The procedure of recruiting participants will be the same in both conditions. The professionals will explicitly invite youths (and their parents) to participate in research with the aim to improve the quality of the Halt-intervention. This will be done (a) verbally during the preliminary conversation, and (b) by sending an invitation flyer with core information about the study immediately after the preliminary conversation. If youths and their parent(s) are interested in participating in the study, they can select a QR-code or link which refers them to the correct information video and an informed consent form corresponding to their age category (-15 years, 16+ years, parents). After giving active consent, youths, and parent(s) (from now on referred to as "participants") are directly referred to the first questionnaire. Participants will be instructed to fill out the first questionnaire before their initial meeting. The procedure for the second and third questionnaires will require no further action from the Halt professionals. All questionnaires will be administered in Dutch and will take approximately 30 minutes to complete per time point.

Data collection

Both recruitment and data collection will start in September 2022. Recruitment will stop after 15 months, because researchers strive to complete pre- and post-tests within 18 months. Follow-up measurements can take place up to 24 months after the start of the data collection. Youths and parents will be asked to fill out three questionnaires: before the intervention, 100 days after the start of the intervention, and 6 months after completion of the intervention. Hundred days is used as a point in time for the post-test because Halt strives to complete all interventions within 100 days.

Aside, from data collected via questionnaires, pseudonymised data from Halt's registration system will be securely transferred to the researchers. These data concerns relevant information regarding the youths, as registered by Halt professionals. For example, offense and referral information (type of crime, prior referrals to Halt, and referral organisation) and Halt-intervention characteristics (confession to the crime, parental consent to Halt, number of meetings between Halt professional and adolescent, and parental presence during meetings). In addition, relevant documents, like the Halt-SI and the YIM-document, are extracted from this system. The Halt-SI, which is administered by all Halt professionals, is a risk assessment tool that assesses various dynamic risk factors (e.g., alcohol use, drug use, and impulsivity) and psychosocial problems (e.g., mood and victim of neglect). In the YIM-document, YIM-trained Halt professionals register information regarding the YIM approach (e.g., the reaction of both youths and parents on the explanation of the YIM approach, which materials are used when motivating the YIM approach, the relationship of the youth with the chosen YIM, etc.). These data will be transferred every three months from Halt to the responsible researcher.

(Statistical) analysis plan

To test similarity between conditions, the two groups of Halt professionals (YIM-trained versus not trained in YIM) will be compared on several demographic factors (age, biological sex, gender identity, educational level, number of years of work experience, number of years working at Halt, and registration at the youth quality register), expectancy outcomes and personality. Second, youths will be compared on demographic factors, offense and referral information, prosocial behaviour and psychosocial problems, and dynamic risk factors. If differences are detected between conditions, propensity score matching (PSM) techniques will be used to match participants from the Halt-plus-YIM condition to the participants in the CAU Halt-condition based on the above-mentioned variables.

For the effect analysis on the different outcome variables, as well as for the moderator and mediator analyses, a series of multiple regression analyses (with baseline levels of the outcome variable as covariate, and condition as predictor variable) will be performed. To correct for the clustering of participants within Halt professionals, the regression analyses will be performed in a multilevel model. To control for chance capitalisation, researchers will implement a Benjamini Hochberg False Detection Rate (FDR) for correction on the p-values for the respective outcome tests.

Power analysis and sample size assessment

To assess the sample size per condition for the primary and secondary outcomes, researchers performed an a priori power analysis in G*Power 3.1. To attain a power level of 0.80 with a significance level of α = .05, a total sample size of N = 100 is necessary to detect a small effect size (f = .10) in a linear multiple regression analysis. For moderator and mediator analysis, a larger sample size is required. Schoemann et al. state that "approximately N = 150 participants are required to ensure statistical power is at least 80% for detecting the hypothesized indirect effect". This would be an indication for a sample size of N = 75 participants per condition. To be able to perform PSM techniques to obtain two comparable groups, researchers will include a doubled ratio in both conditions (N =150 per condition).

A small effect size (f = .10) is expected based on prior knowledge. Prior meta-analyses that explored the effects of formal mentoring programs on delinquent behaviour and reoffending revealed small overall effects, both d = .21 (~f =.10). Even though these effect sizes are small, these demonstrated effect sizes are comparable to other interventions aimed at decreasing delinquent behaviour. It is worthwhile to note that small to medium effect sizes were demonstrated for natural mentoring programs, such as the YIM approach, on positive youth outcomes (g = 0.30). These effects were larger as compared to formal mentoring programs (g = 0.21) and simply the presence of a natural mentor (g = 0.22).

Plan for missing data

Researchers will try to minimise the occurrence of missing data. First, the responsibility of inviting participants for the post-test and follow-up test will lie with the researchers. This will be independent from the intervention adolescents receive at Halt. Thus, even if participants discontinue their intervention at Halt, they will still be approach by the researchers for the post-test and follow-up measurements. Second, the researchers designed the study in way that it relates as much as possible to the participating youth. They are asked how they prefer to be approached and the questionnaires can be easily accessed via their smartphones. This also applies to participating parents.

Missing data is quite unavoidable. Researchers will therefore follow the Intention-to-Treat (ITT) principle for handling missing data on post-test and follow-up measurements. This means that researchers will analyse all missing data of participants according to their assigned condition, regardless of whether the intervention was received or completed. Missing data points will be estimated by performing Full Information Maximum Likelihood (FIML) methods. Researchers will take the percentage of missing data in consideration, and patterns of missing data (e.g., missing completely at random).

ELIGIBILITY:
Inclusion Criteria:

* (First) offenders between 12 and 18 years
* Referred to Halt by the police, prosecutor, special investigating officer, or a school attendance officer after committing an offense or crime
* Three or more meetings with the Halt professional

Exclusion Criteria:

* In both conditions "shortened cases" (i.e., cases with less than 3 meeting) will be excluded. In both conditions, Halt professionals are instructed to follow their regular working process. In the experimental condition, however, YIM trained professionals will be instructed to motivate and explain the YIM for cases with 3 or more meetings. Because motivation and explanation of the YIM approach are usually performed during a follow-up meeting, it will not be possible to motivate and deploy the YIM approach in shortened cases. Therefore, in both conditions, these cases will be excluded from the study.

Ages: 12 Years to 18 Years | Sex: All | Healthy Volunteers: No
Age Groups: Child, Adult
Enrollment: 300 (Estimated)
Dates: Start 2022-09-13 (Actual); Primary Completion 2024-02 (Estimated); Study Completion 2024-08 (Estimated)

PRIMARY OUTCOMES:
Perceived Social Support | Change from baseline at 100 days (post-test)
  Informant: Youth. As measured by the Berlin Social Support Scales (BSSS; Schwarzer & Schulz, 2000): subscale perceived social support. Factor contributing to youth resilience.
Social Resourcefulness | Change from baseline at 100 days (post-test)
  Informant: Youth. As measured by the BSSS (Schwarzer & Schulz, 2000): subscale support seeking. Factor contributing to youth resilience.

SECONDARY OUTCOMES:
Need for (formal) support | Change from baseline at 100 days (post-test)
  Informant: Youth. As measured by the BSSS (Schwarzer & Schulz, 2000): subscale need for support and items from Halt research (Ferwerda et al., 2006). These two scores will be combined to report the youth's need for (formal) support.
Need for (formal) support | Change from baseline at 9 months (follow-up)
  Informant: Youth. As measured by the BSSS (Schwarzer & Schulz, 2000): subscale need for support and items from Halt research (Ferwerda et al., 2006). These two scores will be combined to report the youth's need for (formal) support.
Self-reported delinquency | Change from baseline at 100 days (post-test)
  Informant: Youth. As measured by the Ad Health Self-Reported Delinquency (AHSRD)
Self-reported delinquency | Change from baseline at 9 months (follow-up)
  Informant: Youth. As measured by the Ad Health Self-Reported Delinquency.

OTHER OUTCOMES:
Perceived Social Support | Change from baseline at 9 months (follow-up)
  Informant: Youth. As measured by the Berlin Social Support Scales (BSSS; Schwarzer & Schulz, 2000): subscale perceived social support. Factor contributing to youth resilience.
Perceived Mattering | Change from baseline at 100 days (post-test)
  Informant: Youth. As measured by the General Mattering Scale (GMS; Marcus, 1991). Factor contributing to youth resilience.
Perceived Mattering | Change from baseline at 9 months (follow-up)
  Informant: Youth. As measured by the General Mattering Scale (GMS; Marcus, 1991). Factor contributing to youth resilience.
Relatedness to Others | Change from baseline at 100 days (post-test)
  Informant: Youth. As measured by the Basic Psychological Needs Scale for Adolescents (BPNS-A; Girelli et al., 2019): subscale need for relatedness to others. This adolescent version is adapted from the BPNS of Deci and Ryan (2000). Factor contributing to youth resilience.
Relatedness to Others | Change from baseline at 9 months (follow-up)
  Informant: Youth. As measured by the Basic Psychological Needs Scale for Adolescents (BPNS-A; Girelli et al., 2019): subscale need for relatedness to others. This adolescent version is adapted from the BPNS of Deci and Ryan (2000). Factor contributing to youth resilience.
Peer Network Quality | Change from baseline at 100 days (post-test)
  Informant: Youth. As measured by items on "Delinquent Friends" and "Spending Time with Friends" from the Dutch Research and Documentation Centre (WODC).
Peer Network Quality | Change from baseline at 9 months (follow-up)
  Informant: Youth. As measured by items on "Delinquent Friends" and "Spending Time with Friends" from the Dutch Research and Documentation Centre (WODC).
Social Resourcefulness | Change from baseline at 9 months (follow-up)
  Informant: Youth. As measured by the BSSS (Schwarzer & Schulz, 2000): subscale support seeking. Factor contributing to youth resilience.
Mentor Relationship Quality: Relationship processes | Measured at 100 days
  Informant: Youths. As measured by single items on the type of relationship, frequency of contact, type of activities shared with mentors, duration of the relationship, reliability of the YIM, involvement of parents in choice YIM, and acceptance of choice YIM by parents.
Mentor Relationship Quality: Relationship processes | Measured at 9 months
  Informant: Youths. As measured by single items on frequency of contact, type of activities shared with mentors, duration of the relationship.
Mentor Relationship Quality: Strength of Relationship | Measured at 100 days
  Informant: Youths. As measured by the Youth Strength of Relationship Scale (YSoR): subscale positive. This measurement will be adjusted to measure the youth's perception of the relationship with their YIM.
Mentor Relationship Quality: Strength of Relationship | Change from 100 days at 9 months
  Informant: Youths. As measured by the Youth Strength of Relationship Scale (YSoR): subscale positive. This measurement will be adjusted to measure the youth's perception of the relationship with their YIM.
Competence | Change from baseline at 100 days (post-test)
  Informant: Youth. As measured by the Basic Psychological Needs Scale for Adolescents (BPNS-A; Girelli et al., 2019): subscale need for competence. This adolescent version is adapted from the BPNS of Deci and Ryan (2000). Factor contributing to youth resilience.
Competence | Change from baseline at 9 months (follow-up)
  Informant: Youth. As measured by the Basic Psychological Needs Scale for Adolescents (BPNS-A; Girelli et al., 2019): subscale need for competence. This adolescent version is adapted from the BPNS of Deci and Ryan (2000). Factor contributing to youth resilience.
Autonomy | Change from baseline at 100 days (post-test)
  Informant: Youth. As measured by the Basic Psychological Needs Scale for Adolescents (BPNS-A; Girelli et al., 2019): subscale need for autonomy. This adolescent version is adapted from the BPNS of Deci and Ryan (2000). Factor contributing to youth resilience.
Autonomy | Change from baseline at 9 months (follow-up)
  Informant: Youth. As measured by the Basic Psychological Needs Scale for Adolescents (BPNS-A; Girelli et al., 2019): subscale need for autonomy. This adolescent version is adapted from the BPNS of Deci and Ryan (2000). Factor contributing to youth resilience.
Attitudes towards Delinquency | Change from baseline at 100 days (post-test)
  Informant: Youth. As measured by the Dutch version of the How I Think Questionnaire (HIT-Q; Brugman et al., 2011): subscales on cognitive biases. Factor contributing to youth resilience.
Attitudes towards Delinquency | Change from baseline at 9 months (follow-up)
  Informant: Youth. As measured by the Dutch version of the How I Think Questionnaire (HIT-Q; Brugman et al., 2011): subscales on cognitive biases. Factor contributing to youth resilience.
Parental Monitoring | Change from baseline at 100 days (post-test)
  Informant: Youth. As measured by the Parental Monitoring Scales (PMS; Kerr & Stattin, 2000): subscales Adolescent Disclosure and Parental Solicitation.
Parental Monitoring | Change from baseline at 9 months (follow-up)
  Informant: Youth. As measured by the Parental Monitoring Scales (PMS; Kerr & Stattin, 2000): subscales Adolescent Disclosure and Parental Solicitation.
Attachment to school | Change from baseline at 100 days (post-test)
  Informant: Youth. As measured by the School Connectedness Scale (SCS; Hendrickson Lohmeier & Lee, 2011) and items "Relationship to school" from the Dutch Research and Documentation Centre (WODC).
  Items only relevant if an adolescent goes to school. Factor contributing to youth resilience.
Attachment to school | Change from baseline at 9 months (follow-up)
  Informant: Youth. As measured by the School Connectedness Scale (SCS; Hendrickson Lohmeier & Lee, 2011) and items "Relationship to school" from the Dutch Research and Documentation Centre (WODC).
  Items only relevant if an adolescent goes to school. Factor contributing to youth resilience.
Attachment to work | Change from baseline at 100 days (post-test)
  Informant: Youth. As measured by items "Relationship to work" from the Dutch Research and Documentation Centre (WODC).
  Items only relevant if an adolescent has work. Factor contributing to youth resilience.
Attachment to work | Change from baseline at 9 months (follow-up)
  Informant: Youth. As measured by items "Relationship to work" from the Dutch Research and Documentation Centre (WODC).
  Items only relevant if an adolescent has work. Factor contributing to youth resilience.
Structured free-time activities | Change from baseline at 100 days (post-test)
  Informant: Youth. As measured by items "Free-time activities" from the Netherlands Institute for the Study of Crime and Law Enforcement (NSCR). Factor contributing to youth resilience.
Structured free-time activities | Change from baseline at 9 months (follow-up)
  Informant: Youth. As measured by items "Free-time activities" from the Netherlands Institute for the Study of Crime and Law Enforcement (NSCR). Factor contributing to youth resilience.
Psychosocial Problems | Baseline
  Informant: Youth. As measured by the Dutch version of the Strengths and Difficulties Questionnaire (SDQ; Treffers et al., 2000): subscales emotional problems, behavioural problems, hyperactivity/inattention, and problems with peers.
Prosocial Behaviour | Change from baseline at 100 days (post-test)
  Informant: Youth. As measured by the Dutch version of the Strengths and Difficulties Questionnaire (SDQ; Treffers et al., 2000): subscale prosocial behaviour.
Prosocial Behaviour | Change from baseline at 9 months (follow-up)
  Informant: Youth. As measured by the Dutch version of the Strengths and Difficulties Questionnaire (SDQ; Treffers et al., 2000): subscale prosocial behaviour.
Family Resilience | Change from baseline at 100 days (post-test)
  Informant: Parent(s). As measured by the Family Empowerment Scale (FES; Segers et al., 2019).
Family Resilience | Change from baseline at 9 months (follow-up)
  Informant: Parent(s). As measured by the Family Empowerment Scale (FES; Segers et al., 2019).
Perceived Social Support (Parent(s)) | Change from baseline at 100 days (post-test)
  Informant: Parent(s). As measured by the Berlin Social Support Scales (BSSS; Schwarzer & Schulz, 2000): subscale perceived social support.
Perceived Social Support (Parent(s)) | Change from baseline at 9 months (follow-up)
  Informant: Parent(s). As measured by the Berlin Social Support Scales (BSSS; Schwarzer & Schulz, 2000): subscale perceived social support.
Social Resourcefulness (Parent(s)) | Change from baseline at 100 days (post-test)
  Informant: Parent(s). As measured by the BSSS (Schwarzer & Schulz, 2000): subscale support seeking.
Social Resourcefulness (Parent(s)) | Change from baseline at 9 months (follow-up)
  Informant: Parent(s). As measured by the BSSS (Schwarzer & Schulz, 2000): subscale support seeking.
Parental Stress | Change from baseline at 100 days (post-test)
  Informant: Parent(s). As measured by the Parental Stress Scales (PSS; Berry & Jones, 1995).
Parental Stress | Change from baseline at 9 months (follow-up)
  Informant: Parent(s). As measured by the Parental Stress Scales (PSS; Berry & Jones, 1995).
Parental Monitoring (Parent(s)) | Change from baseline at 100 days (post-test)
  Informant: Parent(s). As measured by the Parental Monitoring Scales (PMS; Kerr & Stattin, 2000): subscales Adolescent Disclosure and Parental Solicitation.
Parental Monitoring (Parent(s)) | Change from baseline at 9 months (follow-up)
  Informant: Parent(s). As measured by the Parental Monitoring Scales (PMS; Kerr & Stattin, 2000): subscales Adolescent Disclosure and Parental Solicitation.
Parent-YIM relationship: Relationship Processes | Measured at 100 days
  Informant: Parent(s). Measured by single items on frequency of contact with YIM, type of relationship with YIM, involvement in the choice of the YIM, acceptance of chosen YIM (whether or not the chosen YIM was agreed upon), and change in relationship with YIM after involvement.
Parent-YIM relationship: Relationship Processes | Change from 100 days measurement at 9 months
  Informant: Parent(s). Measured by single items on frequency of contact with YIM, involvement in the choice of the YIM, acceptance of chosen YIM, and change in relationship with YIM after involvement.
Parent-YIM relationship: Strength of Relationship | Measured at 100 days
  Informant: Youths. As measured by the Youth Strength of Relationship Scale (YSoR): subscale positive. This measurement will be adjusted to measure the parents's perception of the relationship with their YIM.
Parent-YIM relationship: Strength of Relationship | Change from 100 days at 9 months
  Informant: Youths. As measured by the Youth Strength of Relationship Scale (YSoR): subscale positive. This measurement will be adjusted to measure the parents's perception of the relationship with their YIM.
Need for (formal) support (Parent(s)) | Change from baseline at 100 days (post-test)
  Informant: Parent(s). As measured by the BSSS (Schwarzer & Schulz, 2000): subscale need for support and items from Halt research (Ferwerda et al., 2006). These two scores will be combined to report need for formal support.
Need for (formal) support (Parent(s)) | Change from baseline at 9 months (follow-up)
  Informant: Parent(s). As measured by the BSSS (Schwarzer & Schulz, 2000): subscale need for support and items from Halt research (Ferwerda et al., 2006). These two scores will be combined to report need for formal support.
Youth Delinquent Behaviour | Change from baseline at 100 days (post-test)
  Informant: Parent(s). As measured by the Dutch version of the Child Behavior Checklist (CBCL; Verhulst et al., 1997): subscale delinquent behavior.
Youth Delinquent Behaviour | Change from baseline at 9 months (follow-up)
  Informant: Parent(s). As measured by the Dutch version of the Child Behavior Checklist (CBCL; Verhulst et al., 1997): subscale delinquent behavior.

CONTACTS AND LOCATIONS:
Overall Officials: Levi Van Dam, Dr., Principal Investigator — University of Amsterdam; Geertjan J Overbeek, Prof. Dr., Study Director — University of Amsterdam
Locations (1):
- Halt, Utrecht, Netherlands

IPD SHARING:
Plan to Share IPD: Yes
All IPD that underlie results for publication can be made available upon request.
Supporting Information: Study Protocol, ICF
Time Frame: Data will be made available on embargo, three months after the end of the project. This embargo allows researchers to complete ongoing reports on the data, and to take the initiative to develop new publication plans on the project data.
Access Criteria: Via UvA Figshare data can be stored and shared on request. Requests are considered by the study officials. Together they will decide whether anonymised data can be shared with a third party. Files will receive a DOI number, which can be used in articles and presentations.

REFERENCES:
- [Background] Agresti A, Franklin, C. Statistics: The art and science of learning from data. Pearson Education UK; 2013.
- [Background] Benjamini Y, Hochberg, Y. Controlling the false discovery rate: A practical and powerful approach to multiple testing. J R Stat Soc Series B Stat Methodol. 1995;57(1):289-300. https://doi.org/10.1111/j.2517-6161.1995.tb02031.x
- [Background] Bennett DA. How can I deal with missing data in my study? Aust N Z J Public Health. 2001 Oct;25(5):464-9. PMID 11688629
- [Background] Berry J, Jones W. The parental stress scale: Initial psychometric evidence. JSPR. 1995 Aug;12(3):463-472. https://doi.org/10.1177/0265407595123009
- [Background] Bowers EP, Johnson SK, Warren DJA, Tirrel, JM, Lerner JV. Youth-adult relationships and positive youth development. In: Bowers E, Geldhof GJ, editors. Promoting positive youth development. Berlin: Springer; 2015. p. 97-120. https://doi.org/10.1007/978-3-319-17166-1_6
- [Background] Brown, SR. Political subjectivity: Application of Q methodology in political science. New Haven, CT: Yale University; 1980.
- [Background] Brugman D, Nas CN, Van der Velden F, Barriga AQ, Gibbs JC, Bud Potter G, Liau AK. Hoe Ik Denk Vragenlijst (HID): Handleiding (Nederlandse versie). Amsterdam: Boom test uitgevers; 2011.
- [Background] Caliendo M, Kopeinig S. Some practical guidance for the implementation of propensity scoring matching. J Econ Surv. 2008 Jan;22(1):31-72. https://doi.org/10.1111/j.1467-6419.2007.00527.x
- [Background] Deci EL, Ryan, RM. The "what" and "why" of goal pursuits: Human needs and the selfdetermination of behavior. Psychol Inq. 2000 Nov;11:227-268. https://doi.org/10.1207/S15327965PLI1104_01
- [Background] Detry MA, Lewis RJ. The intention-to-treat principle: how to assess the true effect of choosing a medical treatment. JAMA. 2014 Jul 2;312(1):85-6. doi: 10.1001/jama.2014.7523. No abstract available. PMID 25058221
- [Background] DuBois DL, Holloway BE, Valentine JC, Cooper H. Effectiveness of mentoring programs for youth: a meta-analytic review. Am J Community Psychol. 2002 Apr;30(2):157-97. doi: 10.1023/A:1014628810714. PMID 12002242
- [Background] Faul F, Erdfelder E, Buchner A, Lang AG. Statistical power analyses using G*Power 3.1: tests for correlation and regression analyses. Behav Res Methods. 2009 Nov;41(4):1149-60. doi: 10.3758/BRM.41.4.1149. PMID 19897823
- [Background] Ferwerda H, Van Leiden I, Arts N, Hauber A. Halt: Het alternatief? De effecten van Halt beschreven. Advies- en Onderzoeksgroep Beke; Den Haag: Boom Juridische Uitgevers [WODC 'Onderzoek en beleid', nr. 244]; 2006. Retrieved from https://www.researchgate.net/publication/262720839_Halt_Het_Alternatief_De_effecten_van_Halt_beschreven
- [Background] Girelli L, Cavicchiolo E, Lucidi F, Cozzolino M, Alivernini F, Manganelli S. Psychometric properties and validity of a brief scale measuring Basic Psychological Needs Satisfaction in Adolescents. J Educ Cult Psychol Stud. 2019;20:215-229. https://doi.org/10.7358/ecps-2019-020-gire
- [Background] Greeson JK, Usher L, Grinstein-Weiss M. One Adult Who Is Crazy about You: Can Natural Mentoring Relationships Increase Assets among Young Adults With and Without Foster Care Experience? Child Youth Serv Rev. 2010 Apr 1;32(4):565-577. doi: 10.1016/j.childyouth.2009.12.003. PMID 24944430
- [Background] Grollnick WS, Deci EL, Ryan RM. Internalization within the family: The self-determination theory perspective. In: Grusec JE, Kuczynski L, editors. Parenting and children's internalization of values: A handbook of contemporary theory. Hoboken, New Jersey: John Wiley & Sons; 1997. p. 135-161. Retrieved from https://selfdeterminationtheory.org/wp-content/uploads/2020/10/1997_GrolnickDeciRyan.pdf
- [Background] Guest G, Bunce A, Johnson L. How many interviews are enough? An experiment with data saturation and variability. Fields Methods. 2006 Febr;18(1):59-82. https://doi.org/10.1177/1525822X05279903
- [Background] Hawkins S, Karcher MJ, Stewart K, DuBois DL. Mentoring for preventing and reducing delinquent behavior among youth. NMRC Research Review [A Program of Office of Juvenile Justice and Delinquency Prevention]. 2020:1-47. Retrieved from https://nationalmentoringresourcecenter.org/wp-content/uploads/2021/03/Mentoring_for_Preventing_and_Reducing_Delinquent_Behavior_Among_Youth_Research_Review.pdf
- [Background] Hendrickson Lohmeier J, Lee S. A school connectedness scale for use with adolescents. Educational Research and Evaluation. 2011 Apr;12(2):85-95. https://doi.org/10.1080/13803611.2011.597108
- [Background] Jolliffe D, Farrington DP. A rapid evidence assessment of the impact of mentoring on re-offending: A summary [Home Office: Online Report]; 2007 Jul:1-13. Retrieved from https://www.youthmentoring.org.nz/content/docs/Home_Office_Impact_of_mentoring.pdf
- [Background] Kerr M, Stattin H. What parents know, how they know it, and several forms of adolescent adjustment: further support for a reinterpretation of monitoring. Dev Psychol. 2000 May;36(3):366-80. PMID 10830980
- [Background] Marcus, FM. Mattering: Its measurement and theoretical significance for social psychology Cincinnati, OH; 1991.
- [Background] Raposa EB, Rhodes J, Stams GJJM, Card N, Burton S, Schwartz S, Sykes LAY, Kanchewa S, Kupersmidt J, Hussain S. The Effects of Youth Mentoring Programs: A Meta-analysis of Outcome Studies. J Youth Adolesc. 2019 Mar;48(3):423-443. doi: 10.1007/s10964-019-00982-8. Epub 2019 Jan 19. PMID 30661211
- [Background] Schoemann AM, Boulton AJ, Short SD. Determining power and sample size for simple and complex mediation models. Soc Psychol Personal Sci. 2019 Jun;8(4):379-386. https://doi.org/10.1177/1948550617715068
- [Background] Schulz KF, Grimes DA. Sample size slippages in randomised trials: exclusions and the lost and wayward. Lancet. 2002 Mar 2;359(9308):781-5. doi: 10.1016/S0140-6736(02)07882-0. PMID 11888606
- [Background] Schwartz SE, Rhodes JE, Spencer R, Grossman JB. Youth initiated mentoring: investigating a new approach to working with vulnerable adolescents. Am J Community Psychol. 2013 Sep;52(1-2):155-69. doi: 10.1007/s10464-013-9585-3. PMID 23780477
- [Background] Schwarzer R, Schulz U. Berlin Social Support Scales (BSSS). Measurement Instrument Database for the Social Science; 2000. Retrieved from http://userpage.fu-berlin.de/~health/bsss.htm
- [Background] Segers EW, van den Hoogen A, van Eerden IC, Hafsteinsdottir T, Ketelaar M. Perspectives of parents and nurses on the content validity of the Family Empowerment Scale for parents of children with a chronic condition: A mixed-methods study. Child Care Health Dev. 2019 Jan;45(1):111-120. doi: 10.1111/cch.12629. PMID 30426545
- [Background] Tolan PH, Henry DB, Schoeny MS, Lovegrove P, Nichols E. Mentoring Programs to Affect Delinquency and Associated Outcomes of Youth At-Risk: A Comprehensive Meta-Analytic Review. J Exp Criminol. 2014 Jun 1;10(2):179-206. doi: 10.1007/s11292-013-9181-4. PMID 25386111
- [Background] van Dam L, Blom D, Kara E, Assink M, Stams GJ, Schwartz S, Rhodes J. Youth Initiated Mentoring: A Meta-analytic Study of a Hybrid Approach to Youth Mentoring. J Youth Adolesc. 2021 Feb;50(2):219-230. doi: 10.1007/s10964-020-01336-5. Epub 2020 Oct 29. PMID 33123946
- [Background] Van Dam L, Schwartz S. Cultivation of natural mentors to strengthen resilience in youth: A program theory of Youth Initiated Mentoring (YIM). JSI. 2020 Feb;29(1):3-20. https://doi.org/10.18352/jsi.623
- [Background] Van Dam L, Smit D, Wildschut B, Branje SJT, Rhodes JE, Assink M, Stams GJJM. Does Natural Mentoring Matter? A Multilevel Meta-analysis on the Association Between Natural Mentoring and Youth Outcomes. Am J Community Psychol. 2018 Sep;62(1-2):203-220. doi: 10.1002/ajcp.12248. Epub 2018 Apr 25. PMID 29691865
- [Background] Van Dam L, Verhulst S. De JIM-aanpak: Het alternatief voor uithuisplaatsing van jongeren. Amsterdam: Boom Uitgevers; 2018.
- [Background] Van der Laan AM, Blom M. WODC-monitor zelfgerapporteerde jeugdcriminaliteit - meting 2005 [Dutch Research and Documentation Centre]; 2006. Retrieved from https://repository.wodc.nl/bitstream/handle/20.500.12832/882/me2006-4-volledige-tekst_tcm28-67990.pdf?sequence=1&isAllowed=y
- [Background] Verhulst FC, van der Ende J, Koot HM. Handleiding voor de CBCL/4-18. Rotterdam, The Netherlands: Afdeling Kinder- en jeugdpsychiatrie, Sophia Kinderziekenhuis/Academisch Ziekenhuis Rotterdam/Erasmus Universiteit Rotterdam; 1997.
- [Background] Yeatts SD, Martin RH. What is missing from my missing data plan? Stroke. 2015 Jun;46(6):e130-2. doi: 10.1161/STROKEAHA.115.007984. Epub 2015 May 7. No abstract available. PMID 25953373
- [Background] Rhodes JE, Schwartz SEO, Willis MM, Wu MB. Validating a mentoring relationship quality scale: Does match strength predict match length? Youth Soc. 2017 May;49(4): 415-437. https://doi.org/10.1177/0044118X14531604
- [Derived] Boering A, Groenman AP, van Dam L, Overbeek G. Boosters and Barriers to Implementation: Youth-Initiated Mentoring for Justice-Involved Youth. J Community Psychol. 2025 Nov;53(8):e70051. doi: 10.1002/jcop.70051. PMID 41139386
- [Derived] Boering A, Groenman AP, van Dam L, Overbeek G. Effectiveness, working mechanisms, and implementation of youth-initiated mentoring for juvenile delinquents: a multiple-methods study protocol. Health Justice. 2024 Feb 15;12(1):5. doi: 10.1186/s40352-024-00258-9. PMID 38355837